CLINICAL TRIAL: NCT01045902
Title: Prospective, Multi-center, Randomized, Non-blind Trial to Assess the Efficacy and Safety of Moxifloxacin Versus Sulbactam/Ampicillin in the Treatment of Pulmonary Abscess and Aspiration Pneumonia
Brief Title: BAY12-8039, iv/Oral Pulmonary Abscess/Aspiration Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10381
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Pneumonia, Aspiration; Lung Abscess
Keywords: Pulmonary Abscess; Aspiration Pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration; Lung Abscess | interventions — Moxifloxacin; sultamicillin

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)
- Arm 2 (Active Comparator)
  Interventions: Drug: Sulbactam/Ampicillin

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Moxifloxacin, 400 mg iv, od, switch after 6 doses (6 days) to 400 mg Moxifloxacin oral, od
  Arms: Arm 1
Drug: Sulbactam/Ampicillin — Sulbactam/Ampicillin, 3 g iv, tid, switch after 18 doses (6 days) to 750 mg Sulbactam/Ampicillin oral, bid
  Arms: Arm 2

SUMMARY:
The purpose of this trial is to determine the efficacy and safety of Moxifloxacin in comparison to Sulbactam/Ampicillin in the treatment of pulmonary abscesses and aspiration pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or above
* The primary diagnosis is community or hospital acquired primary pulmonary abscess or aspiration pneumonia, requiring initial parenteral treatment

Exclusion Criteria:

* Known hypersensitivity to fluoroquinolones and/or ß-lactams
* Patients with mechanical ventilation lasting more than 48 hours prior to enrollment, with poststenotic pneumonia, infarction pneumonia, pulmonary tuberculosis, lung abscess/pneumonia with concomitant endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2001-02; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Adverse events occuring after first application of study medication up to the test of cure visit for non-serious adverse events | Up to 30 days after end of treatment with study medication for serious adverse events

SECONDARY OUTCOMES:
Clinical Response | Regulary doing i.v. treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- Germany (14):
  - Mannheim, Baden-Wurttemberg
  - Nuremberg, Bavaria
  - Regensburg, Bavaria
  - Treuenbrietzen, Brandenburg
  - Frankfurt am Main, Hesse
  - Hildesheim, Lower Saxony
  - Rotenburg (Wümme), Lower Saxony
  - Lüdenscheid, North Rhine-Westphalia
  - Oberhausen, North Rhine-Westphalia
  - Paderborn, North Rhine-Westphalia
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Lübeck, Schleswig-Holstein
  - Berlin, State of Berlin